CLINICAL TRIAL: NCT02110758
Title: Evaluating the Impact of Patient-Centered Oncology Care
Status: Completed | Type: Observational
Sponsor: National Committee for Quality Assurance (Other)
Collaborators: American Society of Clinical Oncology (Other); Independence Blue Cross (Other); National Coalition for Cancer Survivorship (Unknown); Oncology Management Services (Unknown); RAND (Other)
Responsible Party: Sponsor
Other Study IDs: IH-12-11-4383
Record Dates: First submitted 2014-01-31; First posted 2014-04-10 (Estimated); Results first posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Neoplasms
Keywords: Patient Care Management; Patient Care Planning; Patient-Centered Care; Patient Care Team; Advance Care Planning; Delivery of Health Care; Evidence-based Practice; Health Care Costs; Health Care Quality, Access, and Evaluation; Quality of Health Care; Neoplasms; Medical Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Pilot Practices Patient Survey Cohort: Patients with any active drug therapy treatment for cancer receiving care at pilot practice in southeastern Pennsylvania
  Interventions: Other: Pilot of Patient-Centered Oncology Care
- Comparison Practices Patient Survey Cohort: Patients with any active drug therapy treatment for cancer receiving care at comparison practice in southeastern Pennsylvania
- Pilot Practices Utilization Cohort: Patients with an evaluation & management claim attributed to a medical oncology pilot practice in southeastern Pennsylvania
  Interventions: Other: Pilot of Patient-Centered Oncology Care
- Comparison Practices Utilization Cohort: Patients with an evaluation & management claim attributed to a medical oncology comparison practice in southeastern Pennsylvania
- Pilot Practices Quality Measures Cohort: Patients with a new diagnosis of cancer in the past two years
  Interventions: Other: Pilot of Patient-Centered Oncology Care

INTERVENTIONS:
Other: Pilot of Patient-Centered Oncology Care — Patient-Centered Oncology Care addresses six domains: track & coordinate referrals, provide access and communication, identify and coordinate patient populations, plan and manage care, track & coordinate care, and measure and improve performance.
  Groups: Pilot Practices Patient Survey Cohort; Pilot Practices Quality Measures Cohort; Pilot Practices Utilization Cohort

SUMMARY:
The National Committee for Quality Assurance has worked with the National Coalition for Cancer Survivorship, the American Society of Clinical Oncology, Oncology Management Services, Independence Blue Cross, and RAND, as well as a broader multi-stakeholder advisory group, to define the Patient-Centered Oncology Care model. The purpose of this project was to pilot and evaluate this model. Specific research questions were:

1. Does Patient-Centered Oncology Care improve patient experiences and quality of care? Does it reduce undesirable events like emergency department visits and hospital stays?
2. How does adoption of Patient-Centered Oncology Care vary across a variety of practices and what factors affect adoption?

The demonstration occurred in oncology practices in southeastern Pennsylvania. Practices received implementation support during the 24-month demonstration period. They were evaluated using patient surveys, quality measures, and measures of emergency department and hospital use. Results from these practices were compared in two ways: 1) with their performance before they became oncology medical homes and 2) with other similar practices.

DETAILED DESCRIPTION:
Background. Advances in cancer treatment mean that a growing number of Americans are living with cancer and experiencing it as a chronic, long-term condition. National panels led by consumers have identified the need for improved cancer care in the areas of communication between providers and patients and their families, care planning, attention to nonmedical needs, care coordination and provision of evidence-based treatment. The patient-centered medical home (PCMH) model of care is being widely adopted as a way to provide accessible, proactive, coordinated care and self-care through primary care practices. During active treatment for cancer, the oncology practice is often the primary setting supporting the patient and coordinating cancer treatment. By implementing the patient-centered medical home model, an innovative oncology practice in Pennsylvania has been able to improve access and reduce emergency department visits and hospitalizations for its patients.

Objectives. Building on these recommendations and experience, the National Committee for Quality Assurance has worked with the National Coalition for Cancer Survivorship, the American Society of Clinical Oncology, Oncology Management Services, Independence Blue Cross, and RAND, as well as a broader multi-stakeholder advisory group, to define the Patient-Centered Oncology Care model. We sought PCORI support to pilot and evaluate this model. Specific research questions were:

1. Does Patient-Centered Oncology Care improve patient experiences and quality of care? Does it reduce undesirable events like emergency department visits and hospital stays?
2. How does adoption of Patient-Centered Oncology Care vary across a variety of practices and what factors affect adoption?

Methods. The demonstration occurred in 5 oncology practices in southeastern Pennsylvania. Practices received implementation support during the 24-month demonstration period. They were evaluated using patient surveys, quality measures, and measures of emergency department and hospital use. Results from these practices were compared in two ways: 1) with their performance before they became oncology medical homes and 2) with other similar practices. Patients, clinicians, and health plan leaders helped design the project, and disseminate results. The project used Patient Centered Outcomes Research Institute (PCORI) resources efficiently by building on ongoing efforts. Our evaluation consisted of a retrospective, pre-post study design with a concurrent non-randomized control group of 18 local practices for the utilization and patient experience outcomes. We used difference-in-difference regression models that accounted for practice-level clustering and used functional forms appropriate to the dependent variables. For quality, we compared baseline and follow-up pilot practice performance to national and regional benchmark performance data.

Patient Outcomes. People with cancer are seeking high quality, coordinated and supportive care. The Patient-Centered Oncology Model has the potential to address current gaps in cancer care.

ELIGIBILITY:
Inclusion Criteria

Patients:

* Diagnosis of cancer
* Receives care at a pilot or comparison oncology practice located in southeastern Pennsylvania that accepts patients with Independence Blue Cross health insurance

Exclusion Criteria:

* Any person that does not meet any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients with cancer who received their cancer care from oncology practices. We attributed patients to the study practices (pilot or comparison practices) based on the plurality of office visits for cancer diagnoses. We used sensitivity analyses to investigate other attribution rules, such as the majority of such office visits.
Sampling Method: Non-Probability Sample
Enrollment: 125250 (Actual)
Dates: Start 2014-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah H Scholle, DrPH, MPH, Principal Investigator — National Committee for Quality Assurance
Locations (1):
- National Committee for Quality Assurance, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We didn't follow patients longitudinally. We analyzed cross-sectional patient samples across our pilot and comparison arms in four different time periods: baseline, start-up, intervention & follow-up. Adding up the cross-sectional samples across the periods and arms equals our total enrollment of 125,250 patients.
Groups:
- Pilot Practices Patient Survey Cohort: Patients with any active drug therapy treatment for cancer receiving care at pilot practice in southeastern Pennsylvania
  Intervention:
  Patient-Centered Oncology Care: Patient-Centered Oncology Care addresses six domains: track & coordinate referrals, provide access and communication, identify and coordinate patient populations, plan and manage care, track & coordinate care, and measure and improve performance.
- Comparison Practices Patient Survey Cohort: Patients with any active drug therapy treatment for cancer receiving care at comparison practice in southeastern Pennsylvania
  Intervention:
  No intervention/Usual care
- Pilot Practices Utilization Cohort: Patients with an evaluation & management claim attributed to a medical oncology pilot practice in southeastern Pennsylvania
  Intervention:
  Patient-Centered Oncology Care: Patient-Centered Oncology Care addresses six domains: track & coordinate referrals, provide access and communication, identify and coordinate patient populations, plan and manage care, track & coordinate care, and measure and improve performance.
- Comparison Practices Utilization Cohort: Patients with an evaluation & management claim attributed to a medical oncology comparison practice in southeastern Pennsylvania
  Intervention: No intervention/Usual care
- Pilot Practices Quality Measures Cohort: Patients with a new diagnosis of cancer in the past two years
  Intervention:
  Patient-Centered Oncology Care: Patient-Centered Oncology Care addresses six domains: track & coordinate referrals, provide access and communication, identify and coordinate patient populations, plan and manage care, track & coordinate care, and measure and improve performance.
Period: Baseline: August 2011-July 2013
Arm/Group | Pilot Practices Patient Survey Cohort | Comparison Practices Patient Survey Cohort | Pilot Practices Utilization Cohort | Comparison Practices Utilization Cohort | Pilot Practices Quality Measures Cohort
Started | 0 | 0 | 9832 | 18994 | 308
Completed (This involved cross-sectional samples of patients; we did not follow individuals longitudinally) | 0 | 0 | 9832 | 18994 | 308
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Start-Up: August 2013-June 2014
Arm/Group | Pilot Practices Patient Survey Cohort | Comparison Practices Patient Survey Cohort | Pilot Practices Utilization Cohort | Comparison Practices Utilization Cohort | Pilot Practices Quality Measures Cohort
Started | 175 | 431 | 8057 | 12883 | 0
Completed (This involved cross-sectional samples of patients; we did not follow individuals longitudinally) | 175 | 431 | 8057 | 12883 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Intervention: July 2014-December 2015
Arm/Group | Pilot Practices Patient Survey Cohort | Comparison Practices Patient Survey Cohort | Pilot Practices Utilization Cohort | Comparison Practices Utilization Cohort | Pilot Practices Quality Measures Cohort
Started | 0 | 0 | 10106 | 33012 | 0
Completed (This involved cross-sectional samples of patients; we did not follow individuals longitudinally) | 0 | 0 | 10106 | 33012 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Follow-Up: January-July 2016
Arm/Group | Pilot Practices Patient Survey Cohort | Comparison Practices Patient Survey Cohort | Pilot Practices Utilization Cohort | Comparison Practices Utilization Cohort | Pilot Practices Quality Measures Cohort
Started | 81 | 179 | 6451 | 24392 | 349
Completed (This involved cross-sectional samples of patients; we did not follow individuals longitudinally) | 81 | 179 | 6451 | 24392 | 349
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pilot Practices Utilization Cohort: Patients with any active drug therapy treatment for cancer receiving care at pilot practice in southeastern Pennsylvania
  Intervention:
  Patient-Centered Oncology Care: Patient-Centered Oncology Care addresses six domains: track & coordinate referrals, provide access and communication, identify and coordinate patient populations, plan and manage care, track & coordinate care, and measure and improve performance.
- Comparison Practices Utilization Cohort: Patients with any active drug therapy treatment for cancer receiving care at comparison practice in southeastern Pennsylvania
  Intervention: No intervention/Usual care
- Total: Total of all reporting groups
Arm/Group | Pilot Practices Patient Survey Cohort | Comparison Practices Patient Survey Cohort | Pilot Practices Utilization Cohort | Comparison Practices Utilization Cohort | Pilot Practices Quality Measures Cohort | Total
Number analyzed (Participants) | 256 | 610 | 34446 | 89281 | 657 | 125250
Age, Customized [Count of Participants; unit: Participants]
  18-24 | 0 | 0 | 344 | 894 | 18 | 1256
  25-54 | 36 | 108 | 11385 | 29812 | 173 | 41514
  55-64 | 83 | 177 | 10564 | 26761 | 180 | 37765
  65-74 | 65 | 141 | 5693 | 14116 | 183 | 20198
  75 and older | 64 | 169 | 6460 | 17698 | 103 | 24494
  Unknown | 8 | 15 | 0 | 0 | 0 | 23
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 153 | 386 | 22004 | 59168 | 338 | 82049
  Male | 95 | 209 | 11992 | 30113 | 319 | 42728
  Unknown | 8 | 15 | 0 | 0 | 0 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 137 | 368 | 24571 | 69766 | 416 | 95258
  Black/African-American | 21 | 34 | 6025 | 12117 | 57 | 18254
  Asian | 7 | 6 | 0 | 0 | 9 | 22
  American Indian/Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian/Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Other | 2 | 5 | 0 | 0 | 7 | 14
  Hispanic/Latino | 4 | 6 | 0 | 0 | 14 | 24
  Unknown | 85 | 190 | 3400 | 89281 | 154 | 93110
Region of Enrollment [Number; unit: participants]
  United States | 256 | 610 | 33996 | 89281 | 657 | 65743

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Experience From Baseline to Follow up
Description: Patient experience survey composite scores were evaluated in the pilot practice group and in the comparison practice group during the intervention period and the follow-up period using a modified version of the cancer CAHPS patient survey.
  We calculated survey composite scores on a 0-100 scale using proportional scoring and the summated rating method based on the CAHPS macro.This method calculates the mean responses to each survey item in the composite, after transforming each response to a 0-100 scale (100 representing the most positive response on any given item response scale; 0 representing the least positive). For example, on a Yes/No response scale, if "Yes" represents the most positive response, then Yes= 100 and No = 0; on an Always/Usually/Sometimes/Never response scale, if "Always" represents the most positive response, then Always = 100, Usually = 67, Sometimes = 33 and Never = 0. A higher score means that practices were rated more positively for care on that item.
Time Frame: At baseline and 24 months follow up
Population: Only the Pilot Practices Patient Survey Cohort and Comparison Practices Patient Survey Cohort were pre-specified to be assessed for this Primary Outcome.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Pilot Practices Patient Survey Cohort | Comparison Practices Patient Survey Cohort
Number analyzed (Participants) | 256 | 610
units on a scale
  Affective Communication Composite-Start-Up: number analyzed (Participants) | 175 | 431
  Affective Communication Composite-Start-Up | 90.1 [87.9 to 99.2] | 90.0 [85.7 to 98.8]
  Affective Communication Composite-Follow-Up: number analyzed (Participants) | 81 | 179
  Affective Communication Composite-Follow-Up | 92.8 [82.1 to 97.4] | 92.4 [63.5 to 100]
  Access Composite-Start-Up: number analyzed (Participants) | 175 | 431
  Access Composite-Start-Up | 92.1 [90.6 to 98.9] | 91.0 [79.8 to 99.6]
  Access Composite-Follow-Up: number analyzed (Participants) | 81 | 179
  Access Composite-Follow-Up | 88.4 [83.4 to 94.4] | 93.6 [78.6 to 100]
  Exchanging Information Composite-Start-Up: number analyzed (Participants) | 175 | 431
  Exchanging Information Composite-Start-Up | 88.1 [83.8 to 97.5] | 89.1 [77.8 to 98.2]
  Exchanging Information Composite-Follow-Up: number analyzed (Participants) | 81 | 179
  Exchanging Information Composite-Follow-Up | 86.0 [84.2 to 91.1] | 89.8 [53.9 to 100]
  Patient Self-Management Composite-Start-Up: number analyzed (Participants) | 175 | 431
  Patient Self-Management Composite-Start-Up | 75.2 [68.5 to 86.5] | 76.3 [20.6 to 88.1]
  Patient Self-Management Composite-Follow-Up: number analyzed (Participants) | 81 | 179
  Patient Self-Management Composite-Follow-Up | 67.9 [59.5 to 74.9] | 68.3 [36.6 to 80.7]
  Shared Decision-Making Composite-Start-Up: number analyzed (Participants) | 175 | 431
  Shared Decision-Making Composite-Start-Up | 76.6 [58.7 to 94.5] | 77.9 [41.4 to 95.2]
  Shared Decision-Making Composite-Follow-Up: number analyzed (Participants) | 81 | 179
  Shared Decision-Making Composite-Follow-Up | 83.3 [80.1 to 87.8] | 79.7 [59.3 to 100]
  Overall Rating-Start-Up: number analyzed (Participants) | 175 | 431
  Overall Rating-Start-Up | 92.9 [92.4 to 99] | 90.1 [76.2 to 100]
  Overall Rating-Follow-Up: number analyzed (Participants) | 81 | 179
  Overall Rating-Follow-Up | 89.8 [82.1 to 97.4] | 94.2 [64.5 to 100]
Statistical Analysis 1: Comparison: Pilot Practices Patient Survey Cohort vs Comparison Practices Patient Survey Cohort; To estimate exposure to the intervention on the Access composite score, we used a difference-in-differences model with fixed effects for practices. The dependent variable was the composite score. The intervention effects were represented by the coefficient estimates for survey time period (pre or post) interacted with status (pilot or comparison); Test type: Other; p = .025, Regression, Logistic
Statistical Analysis 2: Comparison: Pilot Practices Patient Survey Cohort vs Comparison Practices Patient Survey Cohort; To estimate exposure to the intervention on the Affective Communication composite score, we used a difference-in-differences model with fixed effects for practices. The dependent variable was the composite score. The intervention effects were represented by the coefficient estimates for survey time period (pre or post) interacted with status (pilot or comparison); Test type: Other; p = 0.69, Regression, Logistic
Statistical Analysis 3: Comparison: Pilot Practices Patient Survey Cohort vs Comparison Practices Patient Survey Cohort; To estimate exposure to the intervention on the Shared Decision-Making composite score, we used a difference-in-differences model with fixed effects for practices. The dependent variable was the composite score. The intervention effects were represented by the coefficient estimates for survey time period (pre or post) interacted with status (pilot or comparison); Test type: Other; p = .013, Regression, Logistic
Statistical Analysis 4: Comparison: Pilot Practices Patient Survey Cohort vs Comparison Practices Patient Survey Cohort; To estimate exposure to the intervention on the Patient Self-Management composite score, we used a difference-in-differences model with fixed effects for practices. The dependent variable was the composite score. The intervention effects were represented by the coefficient estimates for survey time period (pre or post) interacted with status (pilot or comparison); Test type: Other; p = 0.85, Regression, Logistic
Statistical Analysis 5: Comparison: Pilot Practices Patient Survey Cohort vs Comparison Practices Patient Survey Cohort; To estimate exposure to the intervention on the Exchanging Information composite score, we used a difference-in-differences model with fixed effects for practices. The dependent variable was the composite score. The intervention effects were represented by the coefficient estimates for survey time period (pre or post) interacted with status (pilot or comparison); Test type: Other; p = .013, Regression, Logistic
Statistical Analysis 6: Comparison: Pilot Practices Patient Survey Cohort vs Comparison Practices Patient Survey Cohort; To estimate exposure to the intervention on the Overall Rating of Treatment Team composite score, we used a difference-in-differences model with fixed effects for practices. The dependent variable was the composite score. The intervention effects were represented by the coefficient estimates for survey time period (pre or post) interacted with status (pilot or comparison); Test type: Other; p = .053, Regression, Logistic

2. Primary Outcome: Change in Quality of Care From Baseline to Follow up: Percentage of Patients Receiving Recommended Care
Description: Quality measure performance rates were evaluated in the pilot practice group during the baseline period and the follow-up period. Data were abstracted from medical records for a sample of patients diagnosed with an invasive malignancy within previous 2 years and with at least 2 visits to the practice in the previous six months at baseline and at 36 months follow-up.
Time Frame: Two years prior to baseline and at 36 months follow-up
Population: The pilot practices quality measures cohort were pre-specified to be assessed for this outcome. The pilot practices pulled a sample of patient charts at baseline and follow-up (total of 657 patients). Some patients were eligible for specific measures below and some were not.
Measure: Number; unit: percentage of participants
Groups:
- Pilot Practices Quality Measures Cohort: Patients with a new diagnosis of cancer in the past two years
  Patient-Centered Oncology Care: Patient-Centered Oncology Care addresses six domains: track & coordinate referrals, provide access and communication, identify and coordinate patient populations, plan and manage care, track & coordinate care, and measure and improve performance.
Arm/Group | Pilot Practices Quality Measures Cohort
Number analyzed (Participants) | 657
percentage of participants
  Pain assessed, Baseline: number analyzed (Participants) | 307
  Pain assessed, Baseline | 77.9
  Pain assessed, Follow-Up: number analyzed (Participants) | 349
  Pain assessed, Follow-Up | 95.7
  Pain intensity quantified, Baseline: number analyzed (Participants) | 235
  Pain intensity quantified, Baseline | 74.9
  Pain intensity quantified, Follow-Up: number analyzed (Participants) | 329
  Pain intensity quantified, Follow-Up | 94.6
  Plan of care for moderate/severe pain, Baseline: number analyzed (Participants) | 25
  Plan of care for moderate/severe pain, Baseline | 88.3
  Plan of care for moderate/severe pain, Follow-up: number analyzed (Participants) | 61
  Plan of care for moderate/severe pain, Follow-up | 79.5
  Pain addressed defect-free measure, Baseline: number analyzed (Participants) | 307
  Pain addressed defect-free measure, Baseline | 58.8
  Pain addressed defect-free measure, Follow-up: number analyzed (Participants) | 349
  Pain addressed defect-free measure, Follow-up | 87.3
  Emotional well-being assessed, Baseline: number analyzed (Participants) | 266
  Emotional well-being assessed, Baseline | 42.9
  Emotional well-being assessed, Follow-up: number analyzed (Participants) | 349
  Emotional well-being assessed, Follow-up | 75.8
  Emotional well-being addressed, Baseline: number analyzed (Participants) | 65
  Emotional well-being addressed, Baseline | 92.7
  Emotional well-being addressed, Follow-up: number analyzed (Participants) | 78
  Emotional well-being addressed, Follow-up | 84.5
  Documented plan for chemotherapy, Baseline: number analyzed (Participants) | 278
  Documented plan for chemotherapy, Baseline | 96.4
  Documented plan for chemotherapy, Follow-up: number analyzed (Participants) | 290
  Documented plan for chemotherapy, Follow-up | 93.2
  Chemotherapy intent documented, Baseline: number analyzed (Participants) | 276
  Chemotherapy intent documented, Baseline | 80.3
  Chemotherapy intent documented, Follow-up: number analyzed (Participants) | 290
  Chemotherapy intent documented, Follow-up | 92.8
  Chemotherapy intent discussion w/ patient, Baselil: number analyzed (Participants) | 277
  Chemotherapy intent discussion w/ patient, Baselil | 72.5
  Chemotherapy intent discussion with patient, follo: number analyzed (Participants) | 290
  Chemotherapy intent discussion with patient, follo | 87.1
  Number of chemotherapy cycles documented, Baseline: number analyzed (Participants) | 146
  Number of chemotherapy cycles documented, Baseline | 74.5
  Number of chemotherapy cycles documented, Follow-u: number analyzed (Participants) | 149
  Number of chemotherapy cycles documented, Follow-u | 94.6
  Chemotherapy planning defect-free measur, Baseline: number analyzed (Participants) | 276
  Chemotherapy planning defect-free measur, Baseline | 73.2
  Chemotherapy planning defect-free measu, Follow-up: number analyzed (Participants) | 290
  Chemotherapy planning defect-free measu, Follow-up | 86.0
  Chemotherapy treatment summary completed, Baseline: number analyzed (Participants) | 259
  Chemotherapy treatment summary completed, Baseline | 41.1
  Chemotherapy treatment summary completed, Follow-u: number analyzed (Participants) | 80
  Chemotherapy treatment summary completed, Follow-u | 55.6
  Chemotherapy treatment summary to patient, Baselin: number analyzed (Participants) | 255
  Chemotherapy treatment summary to patient, Baselin | 5.6
  Chemotherapy treatment summary to patient, Follow-: number analyzed (Participants) | 78
  Chemotherapy treatment summary to patient, Follow- | 37.3
  Chemotherapy treatment summary to provider, Basel: number analyzed (Participants) | 256
  Chemotherapy treatment summary to provider, Basel | 5.6
  Chemotherapy treatment summary to provider, Follow: number analyzed (Participants) | 73
  Chemotherapy treatment summary to provider, Follow | 41.6
  Chemotherapy treatment defect-free measur Baselin: number analyzed (Participants) | 45
  Chemotherapy treatment defect-free measur Baselin | 15.4
  Chemotherapy treatment defect-free measur Follow-u: number analyzed (Participants) | 76
  Chemotherapy treatment defect-free measur Follow-u | 34.1
  Tobacco use documented, Baseline: number analyzed (Participants) | 298
  Tobacco use documented, Baseline | 89.7
  Tobacco use documented, Follow-up: number analyzed (Participants) | 343
  Tobacco use documented, Follow-up | 99.6
  Tobacco use cessation recommended, Baseline: number analyzed (Participants) | 38
  Tobacco use cessation recommended, Baseline | 51.6
  Tobacco use cessation recommended, Follow-up: number analyzed (Participants) | 50
  Tobacco use cessation recommended, Follow-up | 47.1
  Tobacco use cessation administered, Baseline: number analyzed (Participants) | 38
  Tobacco use cessation administered, Baseline | 43.5
  Tobacco use cessation administered, Follow-up: number analyzed (Participants) | 50
  Tobacco use cessation administered, Follow-up | 16.7
  Tobacco defect-free measure, Baseline: number analyzed (Participants) | 298
  Tobacco defect-free measure, Baseline | 89.5
  Tobacco defect-free measure, Follow-up: number analyzed (Participants) | 343
  Tobacco defect-free measure, Follow-up | 85.8
  Serotonin antagonist prescribed, Baseline: number analyzed (Participants) | 97
  Serotonin antagonist prescribed, Baseline | 98.5
  Serotonin antagonist prescribed, Follow-up: number analyzed (Participants) | 228
  Serotonin antagonist prescribed, Follow-up | 98.7
  Sertonin antagonist/corticosteroids, Ba: number analyzed (Participants) | 215
  Sertonin antagonist/corticosteroids, Ba | 89.9
  Serotonin antagonist/corticosteroids, Follow-up: number analyzed (Participants) | 228
  Serotonin antagonist/corticosteroids, Follow-up | 88.8
  Aprepitant prescribed, Baseline: number analyzed (Participants) | 101
  Aprepitant prescribed, Baseline | 84.9
  Aprepitant prescribed, Follow-up: number analyzed (Participants) | 72
  Aprepitant prescribed, Follow-up | 75.8
  Anti-emetics defect-free measure, Baseline: number analyzed (Participants) | 214
  Anti-emetics defect-free measure, Baseline | 71.2
  Anti-emetics defect-free measure, Follow-up: number analyzed (Participants) | 129
  Anti-emetics defect-free measure, Follow-up | 92.5
  Infertility risks discussed, Baseline: number analyzed (Participants) | 39
  Infertility risks discussed, Baseline | 28.3
  Infertility risks discussed, Follow-up: number analyzed (Participants) | 28
  Infertility risks discussed, Follow-up | 63.4
  Fertility preservation options discussed, Baseline: number analyzed (Participants) | 39
  Fertility preservation options discussed, Baseline | 52.5
  Fertility preservation options discussed, Follow-u: number analyzed (Participants) | 28
  Fertility preservation options discussed, Follow-u | 63.9

3. Primary Outcome: Change in Health Care Utilization From Baseline to Follow up
Description: Per member per month hospitalizations, emergency department visits, primary care visits and specialist visits were evaluated in the pilot group and in the comparison group using insurance claims data during the baseline, start-up, intervention and follow-up periods.
Time Frame: Two years prior to baseline and at 36 months follow up
Population: Only the Pilot Practices Utilization Cohort and Comparison Practices Utilization Cohort were pre-specified to be assessed for this outcome
Measure: Mean (Full Range); unit: Per member per month visits
Groups:
- Pilot Practices Utilization Cohort: Patients with an evaluation & management claim attributed to a medical oncology pilot practice in southeastern Pennsylvania
  Patient-Centered Oncology Care: Patient-Centered Oncology Care addresses six domains: track & coordinate referrals, provide access and communication, identify and coordinate patient populations, plan and manage care, track & coordinate care, and measure and improve performance.
Arm/Group | Pilot Practices Utilization Cohort | Comparison Practices Utilization Cohort
Number analyzed (Participants) | 34446 | 89281
Per member per month visits
  All-cause hospitalizations, Baseline: number analyzed (Participants) | 9832 | 18994
  All-cause hospitalizations, Baseline | 0.0403 [0 to 0.8750] | 0.0386 [0 to 1.3333]
  All-cause hospitalizations, Start-up: number analyzed (Participants) | 8057 | 12883
  All-cause hospitalizations, Start-up | 0.0484 [0 to 1.6364] | 0.0823 [0 to 1.7273]
  All-cause hospitalizations, Intervention: number analyzed (Participants) | 10106 | 33012
  All-cause hospitalizations, Intervention | 0.0623 [0 to 1.3333] | 0.0512 [0 to 1.1667]
  All-cause hospitalizations, Follow-up: number analyzed (Participants) | 6451 | 24392
  All-cause hospitalizations, Follow-up | 0.0574 [0 to 1.7143] | 0.0529 [0 to 2.2857]
  All-cause ED visits, Baseline: number analyzed (Participants) | 9832 | 18994
  All-cause ED visits, Baseline | 0.0815 [0 to 2.6667] | 0.0781 [0 to 4.1667]
  All-cause ED visits, Start-up: number analyzed (Participants) | 8057 | 12883
  All-cause ED visits, Start-up | 0.0873 [0 to 4.6364] | 0.0973 [0 to 6.0000]
  All-cause ED visits, Intervention: number analyzed (Participants) | 10106 | 33012
  All-cause ED visits, Intervention | 0.0825 [0 to 9.5556] | 0.0833 [0 to 3.2778]
  All-cause ED Visits, Follow-up: number analyzed (Participants) | 6451 | 24392
  All-cause ED Visits, Follow-up | 0.0969 [0 to 3.8571] | 0.1008 [0 to 4.2857]
  PCP Office Visits, Baseline: number analyzed (Participants) | 9832 | 18994
  PCP Office Visits, Baseline | 0.2539 [0 to 3.5417] | 0.2505 [0 to 5.0417]
  PCP Office Visits, Start-Up: number analyzed (Participants) | 8057 | 12883
  PCP Office Visits, Start-Up | 0.2657 [0 to 10.909] | 0.2679 [0 to 8.6364]
  PCP Office Visits, Intervention: number analyzed (Participants) | 10106 | 33012
  PCP Office Visits, Intervention | 0.2764 [0 to 5.0556] | 0.2781 [0 to 12.889]
  PCP Office Visits, Follow-up: number analyzed (Participants) | 6451 | 24392
  PCP Office Visits, Follow-up | 0.2731 [0 to 4.4286] | 0.2731 [0 to 11.857]
  Specialist Office Visits, Baseline: number analyzed (Participants) | 9832 | 18994
  Specialist Office Visits, Baseline | 0.9211 [0 to 18.208] | 0.8967 [0 to 8.7083]
  Specialist Office Visits, Start-Up: number analyzed (Participants) | 8057 | 12883
  Specialist Office Visits, Start-Up | 0.9211 [0 to 18.208] | 0.8967 [0 to 8.7083]
  Specialist Office Visits, Intervention: number analyzed (Participants) | 10106 | 33012
  Specialist Office Visits, Intervention | 1.0199 [0 to 16.545] | 1.0141 [0 to 17.636]
  Specialist Office Visits, Follow-Up: number analyzed (Participants) | 6451 | 24392
  Specialist Office Visits, Follow-Up | 1.0018 [0 to 10.167] | 0.9549 [0 to 11.111]
Statistical Analysis 1: Comparison: Pilot Practices Utilization Cohort vs Comparison Practices Utilization Cohort; To estimate exposure to the intervention on Per Member Per Month Hospitalizations, we used a difference-in-differences model with fixed effects for practices. The dependent variable was Per Member Per Month Hospitalizations. The intervention effects were represented by the coefficient estimates for utilization time period (baseline or follow-up) interacted with status (pilot or comparison); Test type: Other; p = 0.2, Regression, Logistic
Statistical Analysis 2: Comparison: Pilot Practices Utilization Cohort vs Comparison Practices Utilization Cohort; To estimate exposure to the intervention on Per Member Per Month Emergency Department (ED) Visits, we used a difference-in-differences model with fixed effects for practices. The dependent variable was Per Member Per Month ED Visits. The intervention effects were represented by the coefficient estimates for utilization time period (baseline or follow-up) interacted with status (pilot or comparison); Test type: Other; p = 0.62, Regression, Logistic
Statistical Analysis 3: Comparison: Pilot Practices Utilization Cohort vs Comparison Practices Utilization Cohort; To estimate exposure to the intervention on Per Member Per Month Primary Care Visits, we used a difference-in-differences model with fixed effects for practices. The dependent variable was Per Member Per Month Primary Care Visits. The intervention effects were represented by the coefficient estimates for utilization time period (baseline or follow-up) interacted with status (pilot or comparison); Test type: Other; p = 0.68, Regression, Logistic
Statistical Analysis 4: Comparison: Pilot Practices Utilization Cohort vs Comparison Practices Utilization Cohort; To estimate exposure to the intervention on Per Member Per Month Specialist Visits, we used a difference-in-differences model with fixed effects for practices. The dependent variable was Per Member Per Month Specialist Visits. The intervention effects were represented by the coefficient estimates for utilization time period (baseline or follow-up) interacted with status (pilot or comparison); Test type: Other; p = 0.03, Regression, Logistic

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Pilot Practices Patient Survey Cohort | Comparison Practices Patient Survey Cohort | Pilot Practices Utilization Cohort | Comparison Practices Utilization Cohort | Pilot Practices Quality Measures Cohort
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes